CLINICAL TRIAL: NCT07275528
Title: Effects of Task Oriented Circuit Training on Functional Mobility and Activity Participation in Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/10
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy (CP); Functional Mobility
Keywords: Task oriented circuit training; functional mobility; activity participation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- task oriented circuit training (Experimental): Task-oriented circuit training was delivered through a structured set of fourteen workstations designed to promote functional mobility, strength, balance, and coordination. Each workstation targeted a specific task, such as standing and reaching beyond arm's length at various distances and heights, sit-to-stand transitions from different chair heights, multidirectional stepping on blocks of varying heights and surfaces, alternating heel and toe raising, and progressive squatting with adjustments in depth, duration, and added hand weights. Additional stations included supine straight leg raises with optional cuff weights, stair ascending and descending with progressive load, backward walking beginning near a wall and advancing to open space with shuttle runs, walking on a balance beam with speed and surface variations, core-strengthening crunches, supine bridging with increased knee flexion and repetitions, prone opposite arm-and-leg raises with repetition progression, side bridge exer
  Interventions: Procedure: Experimental
- Conventional physical therapy (Other): convention physical therapy will provide to both the groups comprised stretching exercises, strengthening exercises and positioning. Each spastic muscle will stretch up to the level of mild discomfort where it was held for 20 seconds and the procedure was repeated five times. Each CP child will assess separately for spastic group of muscles. Each weak muscle was made to contract against resistance 10 times in one session. Parents will advise to make their child sit with open legs on bench/block with heels touching the ground. They will also advise to make standing position against a wall with legs in moderate abduction and external rotation for 15 minutes daily after exercises
  Interventions: Procedure: CONVENTIONAL PHYSICAL THERAPY

INTERVENTIONS:
Procedure: Experimental — The intervention consists of a structured taskoriented circuit training program composed of 14 different workstations designed to target functional mobility, lower limb strength, balance, and endurance. Each station addresses a specific motor task, such as standing and reaching, sit-to-stand from variable chair heights, multidirectional stepping on firm and soft surfaces, alternating heel-toe raises, progressive squats (with modifications in depth, duration, and added weight), supine straight leg raises, stair climbing (ascending and descending), backward walking, balance beam walking, core strengthening via crunches and bridges, prone alternating arm/leg raises, side bridges, and cycling on a stationary bicycle with adjustable resistance and direction.
  Arms: task oriented circuit training
Procedure: CONVENTIONAL PHYSICAL THERAPY — Sessions: 3 sessions per week (30-40 minutes) Duration: 6-8 weeks Frequency: 3-4 sessions/week Session Length: 30-40 minutes Format: begin with less repetition gradually progress to increase time and repetition HOT PACK: 10 MINS Week 1-2
  1. Stretching Exercises Exercise Detail: Spastic muscles are stretched to the point of mild discomfort. Each stretch is held steadily while maintaining proper alignment. Dosage: Hold each stretch for 20 seconds and repeat 5 times for every identified spastic muscle.
  2. Strengthening Exercises Exercise Detail: Weak muscles are activated through gentle contractions performed against light resistance. Dosage: Perform 10 repetitions for each weak muscle in every session.
  3. Positioning Exercise Detail: Child is positioned in sitting with legs open on a bench or block, heels touching the ground. Standing against a wall with moderate abduction and external rotation is also introduced. Dosage: Maintain sitting as tolerated. Wall -standing for 15 minutes
  Arms: Conventional physical therapy

SUMMARY:
cerebral palsy hemiplegia often experiences motor problems that primarily affect one side of their body. Children with hemiplegia have difficulties in functional activities. Task-Oriented Circuit Training (TOCT) is a high-intensity, progressive intervention designed to improve functional motor skills by engaging individuals in repetitive, task-specific exercis it is randomized control trail conducted with 34 patients included according to inclusion and exclusion criteria. Functional mobility assessed through 6-minute walk test and activity participation evaluated through Child Engagement in Daily Life measurement scale.

DETAILED DESCRIPTION:
Cerebral palsy hemiplegia often experiences motor problems that primarily affect one side of their body. Children with hemiplegia have difficulties in functional activities, which severely affects the children's quality of life. Task-Oriented Circuit Training (TOCT) is a progressive intervention designed to improve functional motor skills by engaging individuals in repetitive, task-specific exercises. It involves a series of workstations where individuals practice tasks like balancing, walking, and reaching skills essential for daily life. The purpose of the research was to find out the effectiveness of task specific circuit training on activity participation and functional mobility in children with hemiplegic cerebral palsy. This non blinded randomized control trail will be conducted at fauji foundation hospital Rawalpindi for the duration of 1 year after approval of GERC with 34 patients included according to inclusion and exclusion criteria. After ethical approval from FUSH ERC, eligible participants will be randomly assigned into two groups through sealed envelope method. The participants would assess through 6- minute walk test for functional mobility and child engagement in daily life measurement scale for activity participation on the day of starting the intervention, after 4th week and 8th week. Intervention will be given for a total 40-50 minutes per session, 3 sessions per week for consecutive 8 weeks. Task-oriented Circuit Training (TSCT) includes 14 workstations that target different motor skills through progressive exercises that gradually increase in difficulty. Conventional Physical Therapy includes Stretching of tight muscles, strengthening of weak muscles, and positioning

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of hemiplegic cerebral palsy
* Both genders are included
* The children were between 5 and 12 years old.
* Their motor function was at a level I or II based on the GMFCS,
* The degree of spasticity grade 1 to 2 based on the Modified Ashworth Scale.

Exclusion Criteria:

* Visual or hearing loss
* Cognitive impairment
* Seizures
* A botulinum toxin injection in the previous six months,
* Lower extremity surgery
* Musculoskeletal disorders
* Structural deformities in the spine and/or lower limbs.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
activity participation | 6 weeks
  activity participation is assessed by child engagement in daily life measurement scale. A CEDL scaled score ranges from 0 to 100, where 100 indicates the highest level of participation or independence, 70-90 suggests moderate participation, 40-60 indicates limited or inconsistent participation, and below 40 represents significant restrictions
Functional mobility | 6 weeks
  functional mobility assessed by 6-minute walk test functional changes were evaluated using the minimal clinically important difference (MCID) reported for children with CP.
  Changes exceeding 6-23 meters is significant. Difference less than 6 meters is insignificant.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan